CLINICAL TRIAL: NCT06229574
Title: The Effect of Antenatal Breastfeeding Education Prepared With Virtual Reality Technology on Breastfeeding Self-Efficacy and Breastfeeding Success of Primiparous Mothers
Brief Title: Breastfeeding Education Prepared With Virtual Reality Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, ipek turhan, nurse, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ErciyesU-SBF-IT-01
Record Dates: First submitted 2023-12-21; First posted 2024-01-29 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Breast Feeding
Keywords: Breast Milk; Breast-feeding; Breastfeeding Education; Virtual Reality
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: The research will be conducted as an experimental single-blind study with a randomized control group.
Who Masked: Outcomes Assessor
Masking Description: The application was administered to the participants by the researcher, but postpartum breastfeeding success and breastfeeding self-efficacy were evaluated by an interviewer who was unaware of the participants' group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): The effect of breastfeeding education given with virtual reality glasses on breastfeeding success and breastfeeding self-efficacy will be evaluated. The education given during pregnancy will be evaluated on the first and seventh days after birth.
  Interventions: Other: virtual reality glasses
- control group (No Intervention): Breastfeeding success and breastfeeding self-efficacy of women included in this group during pregnancy will be evaluated on the first and seventh days after birth.

INTERVENTIONS:
Other: virtual reality glasses — The breastfeeding software developed will be applied in this group.
  Arms: intervention group

SUMMARY:
The breastfeeding software developed with the primiparous study was transferred to virtual reality glasses. This study will be applied to pregnant women and its effect on breastfeeding success and breastfeeding self-efficacy will be investigated.

DETAILED DESCRIPTION:
The goal of this clinical trial is to To learn The Effect Of Pre-Natal Breastfeeding Education Prepared Wıth Virtual Reality Technology On The Breastfeeding Self-Efficiency And Breastfeeding Success Of Primiparous Mothers in The study will be delivered to 60 healthy primiparous pregnant women.The breastfeeding software developed with the primary study was transferred to virtual reality glasses. It will also be implemented in this study. The main questions it aims to answer are:

* Prenatal breastfeeding education prepared with virtual reality technology positively affects the breastfeeding self-efficacy of primiparous mothers.
* Prenatal breastfeeding education prepared with virtual reality technology positively affects the breastfeeding of primiparous mothers.

Participants will Pregnant women in the intervention group will be given breastfeeding training prepared with virtual reality technology and will fill out questionnaires and scales will be filled in on the first and seventh days after birth. Questionnaires will be filled in by pregnant women in the control group, and the scales will be filled out only on the first and seventh days.

Researchers will compare breastfeeding education given with virtual reality glasses with the control group to see whether it has an effect on breastfeeding success and breastfeeding self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 35
* literate,
* Pregnant women who are at 37 weeks of gestation and above,
* Those with healthy pregnancies (singleton pregnancy, no systemic/chronic disease, etc.) -Primiparous pregnant women-
* Vaginal birth planned,
* planning to breastfeed,
* Those who do not have any problems with their breasts that would make breastfeeding difficult (collapsed, missing tip, wound on the nipple, etc.),
* Pregnant women who do not have vision, hearing or communication problems
* Pregnant women who do not have any problems will be included in the study.

Exclusion Criteria:

* Occurrence of a situation that prevents sucking
* Baby with congenital anomalies

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since it is a study on breastfeeding, it is a study specific to women.
Enrollment: 59 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
breastfeeding success | 4-5 week
  LACTH BREASTFEEDING ASSESSMENT SCALE This measurement tool consists of five evaluation criteria and is a combination of the first letters of the English equivalents of these criteria. Each item is evaluated between 0 and 2 points. The total score that can be obtained from the measurement tool is 10. The measurement tool has no cutoff point. It is understood that the higher the LATCH score, the higher the breastfeeding success.
breastfeeding self-efficacy | 4-5 week
  breastfeeding self-efficacy scale The Turkish validity and reliability of the Breastfeeding Self-Efficacy Scale Short Form was conducted by Aluş Tokat and Okumuş in 2009 . This scale evaluates how competent mothers feel regarding breastfeeding. The scale consists of 14 items and includes a 5-point Likert-type evaluation consisting of the options: Not at all sure , Very not sure , Sometimes sure , Sure and Very sure . The lowest score that can be obtained from the entire scale is 14 and the highest score is 70. A high score from the scale indicates a high perception of breastfeeding self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: ipek turhan, master, Principal Investigator — Kayseri City Hospital
Locations (1):
- Ipek Turhan, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No